CLINICAL TRIAL: NCT02253121
Title: Randomized, Double-blind, Placebo-controlled Trial on the Effectiveness and Safety of Dapagliflozin for Blood Glucose Control During Glucocorticoid Treatment for Acute Exacerbation COPD
Brief Title: Glucose Control During Glucocorticoid Therapy in Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: GluCon-COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Slotervaart Hospital (Other)
Collaborators: AstraZeneca (Industry); Isala (Other); Spaarne Gasthuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL49690.048.14; 2014-001877-15 (EudraCT Number)
Record Dates: First submitted 2014-09-22; First posted 2014-10-01 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Hyperglycemia Steroid-induced
Keywords: COPD; acute exacerbation; glucocorticoid therapy; hyperglycemia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hyperglycemia | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin + sliding scale insulin. (Experimental): Treatment with dapagliflozin 10mg once daily orally. Treatment will start as soon as possible after initation of glucocorticoid pulse therapy for acute exacerbation COPD and will end when pulse therapy is finished (expected duration 10-14 days). In case of persistent glucose levels > 12 mmol/l, subjects will receive escape treatment with sliding scale insulin.
  Interventions: Drug: Dapagliflozin; Drug: Sliding scale insulin
- Placebo + sliding scale insulin (Placebo Comparator): Treatment with placebo once daily orally. Treatment will start as soon as possible after initation of glucocorticoid pulse therapy for acute exacerbation COPD and will end when pulse therapy is finished (expected duration 10-14 days). In case of persistent glucose levels > 12 mmol/l, subjects will receive escape treatment with sliding scale insulin.
  Interventions: Drug: Sliding scale insulin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10mg during glucocorticoid therapy for acute exacerbation COPD
  Other Names: Forxiga
  Arms: Dapagliflozin + sliding scale insulin.
Drug: Sliding scale insulin — Sliding scale insulin with short acting insulin based on current glucose levels
  Other Names: Supplemental insulin

SUMMARY:
Purpose of this study is to treat glucocorticoid induced hyperglycemia due to glucocorticoid pulse therapy in a efficacious, safe and convenient way. Patients with acute exacerbation of COPD treated with glucocorticoid pulse therapy and at high risk for glucocorticoid induced hyperglycemia (defined as known type 2 DM or glucose > 10mmol/l at admission) will be randomized to treatment of dapagliflozin or placebo orally, once daily.

Percentage of time within glucose target range (3,9-10 mmol/l) and incidence rate of hypoglycemia will be compared between dapagliflozin group and placebo group.

DETAILED DESCRIPTION:
Rationale: Patients hospitalized for COPD exacerbation treated with high dose glucocorticoids, frequently develop hyperglycaemia. Currently, sliding scale insulin is often used to bridge such episodes. However, sliding scale insulin is patient unfriendly, does not reduce glycaemic excursion nor glycaemic variability. In contrast, pharmacologic inhibition of the sodium glucose transporter-2 (SGLT-2) can be given as an oral agent and is likely to result in better glucose control with lower risk of hypoglycaemia Objective: glucose control and safety (risk of hypoglycaemia). Secondary objectives are patient satisfaction, other safety outcomes and other parameters of glucose control Study design: Double-blind placebo controlled intervention study Study population: Patients hospitalized for an exacerbation of chronic obstructive lung disease who are treated with high dose glucocorticoids.

Intervention: One group receives once daily a 10mg tablet of dapagliflozin and the other group receives once daily a placebo tablet as add on to their prestudy glucose-lowering medication. Both groups will be treated with glucose lowering escape medication if required.

Main study parameters/endpoints: Glucose control is measured as the average time spent within target range in each patient. Safety is measured as the incidence rate of hypoglycaemia during study follow-up.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden of participation consists of the extra capillary glucose measurements that will be done 3-4 times daily and wearing a coin size glucose sensor. Furthermore, patients have to fill out a treatment satisfaction questionnaire. There will be no extra site visits for participants.

Dapagliflozin (experimental group) carries a risk of hypoglycaemia, especially for patient who have concomitant therapy with insulin or sulfonylurea derivatives. Patients will be instructed to anticipate, and if required dosing of glucose lowering therapy will be adjusted. Furthermore, dapagliflozin carries an increased risk of urogenital infections, increased haematocrit and LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Hospitalization due to AECOPD
* Treatment with ≥30mg prednisone daily or equivalent dose of glucocorticoid for AECOPD
* An expected duration of glucocorticoid treatment of 3-14 days at study entry
* Known type 2 diabetes or glucose ≥ 10 mmol/l at admission

Exclusion Criteria:

* High dose glucocorticoid treatment started ≥7 days before study entry
* Need for ICU admission
* Chronic kidney disease stage G3 (glomerular filtration rate <60ml/minute)
* Recurrent genital or urinary tract infection
* Current use of any SGLT-2 inhibiting agent
* Suspected volume depletion
* Congestive heart failure functional classification NYHA class IV/IV or instable heart failure
* Acute stroke within 2 months before inclusion.
* Recent cardiovascular event: acute coronary syndrome, hospitalisation for unstable angina or coronary revascularisation within 2 months before inclusion
* Suspected liver disease, confirmed by AST/ALT > 3x ULN or bilirubin >2.0mg/dl (34.2 μmol/l) or serologically proven infection with hepatitis B or hepatitis C
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Glucose control | 2nd till 7th day of treatment
  % time within target range (3.9-10 mmol/l)
Risk of hypoglycemia | Randomisation till end of study (expected duration of 12 days)
  Incidence rate of hypoglycaemic events

SECONDARY OUTCOMES:
Patient satisfaction | During hospital stay (expected average of 9 days)
  Diabetes treatment satisfaction questionnaire for inpatients
Clinical outcomes | During hospital stay (expected average of 9 days)
  Duration of hospitalisation, need for treatment escalation, incidence (re-)infections, change in body weight and blood pressure.
Safety | Randomisation till end of study (expected duration of 12 days)
  incidence rate of asymptomatic hypoglycaemia, incidence adverse events of special interest (genital infections, urinary tract infections, renal impairment, liver injury and breast-, bladder- and prostate cancer), incidence of other adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Gerdes, MD, PhD, Principal Investigator — Slotervaart Hospital
Locations (4):
- Netherlands (4):
  - Slotervaart Hospital, Amsterdam
  - OLVG West, Amsterdam
  - Spaarne Ziekenhuis, Hoofddorp
  - Isala, Zwolle

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5947126/